CLINICAL TRIAL: NCT03899142
Title: Pharmacokinetics of HepBQuin Manufactured According to a New Production Process
Brief Title: Pharmacokinetics of New HepBQuin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MD2017.01
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- human hepatitis B immunoglobulin (Experimental): once, i.m.
  Interventions: Biological: a human hepatitis B immunoglobulin solution for injection for intramuscular administration

INTERVENTIONS:
Biological: a human hepatitis B immunoglobulin solution for injection for intramuscular administration — intramuscular administration

SUMMARY:
Sanquin Plasma Products BV developed a new manufacturing process for the Quin plasma products in order to improve viral safety and to remove procoagulant activity. Since the new manufacturing process will be the same for all Quin products, a clinical study with one of the Quin products is sufficient for marketing authorisation of all new Quin products. HepBQuin will serve as model for all other Quin products. Pharmacokinetic (PK) data are considered as a surrogate indicator of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male and female, aged 18 to 65 inclusive.
* Negative serology test for HBsAg, anti-HBs, and anti-HBc at screening.
* Body-mass index (BMI) of 18.5 to 32.0 kg/m2 (inclusive).
* Female volunteers must have a pregnancy test at screening.
* Willing to participate by signing the written signed informed consent form.

Exclusion Criteria:

* Vaccinated against Hepatitis B
* Having a Hepatitis B infection or suffered from a Hepatitis B infection in the past.
* Known with allergic reactions against human plasma, plasma products or blood products.
* A history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening.
* Thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Known with or having a history of arterial or venous thromboembolic events.
* Pre-existing risk factors for thrombotic events.
* Any clinically significant history of or current clinically significant other disease or disorder.
* Any clinically significant abnormality following the investigator's review of physical examination, and clinical laboratory tests obtained at screening.
* An abnormal pulse rate and/or blood pressure measurements at the screening visit.
* Pregnant or breast-feeding at screening or at Day 0
* Women of childbearing potential not using a highly effective method of birth.
* Any use of drugs or abuse within 3 months prior to screening and during study.
* Alcohol abuse within 3 months prior to screening and during study
* Participated in another interventional clinical trial a month before the start of the study, or having received an experimental drug during the previous 30 days.
* Having IgA deficiency with anti-IgA antibodies.
* Blood or plasma donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
half-life of anti-HBs antibodies | 84 days
  Pharmacokinetics

SECONDARY OUTCOMES:
number of adverse events | 84 days
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No